CLINICAL TRIAL: NCT03347136
Title: Comparison of CPAP and NIPPV as a Mode of Non-invasive Respiratory Support for Neonates in a Level III NICU
Brief Title: Comparison of Continuous Positive Airway Pressure and Non Invasive Positive Pressure Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Sri Lanka (Other Government)
Responsible Party: Principal Investigator, Dr. Anne kaushalya Shilani Gomez,MBBS,MD, acting consultant neonatologist, Ministry of Health, Sri Lanka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHSriLanka
Record Dates: First submitted 2017-11-10; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Respiratory Distress of Newborn
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: The neonates with mild to moderate respiratory distress were randomly allocated to tratment with NIPPV and CPAP.
Masking Description: Due to type of intervention masking was not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newborns with CPAP support (Active Comparator): Newborn with mild to moderate respiratory distress randomly allocated to CPAP arm. CPAP started with Positive End Expiatory Pressure(PEEEP) 05 and increased up to PEEP 09 according to the severity of baby's condition.
  Interventions: Device: CPAP
- Newborns with NIPPV support (Experimental): Newborn with mild to moderate respiratory distress randomly allocated to NIPPV arm. NIPPV started with Intermittent Mandatory Ventilation rate 30, Peak Inspiratory Pressure 20 and PEEP 5.Increased the settings according to the severity of baby's condition
  Interventions: Device: NIPPV

INTERVENTIONS:
Device: CPAP
  Arms: Newborns with CPAP support
Device: NIPPV
  Arms: Newborns with NIPPV support

SUMMARY:
The objective of the study is to compare the effectiveness of treatment with Non Invasive Positive Pressure Ventilation (NIPPV) and continuous positive airway pressure (CPAP) in decreasing the requirement for endotracheal ventilation in neonates with respiratory distress within the first hours of birth.Primary outcome is the non invasive respiratory support failure and the need for intubated ventilatory support during the first 72 hours of life.

Randomized control , single center trial. Eighty neonates admitted to Neonatal Intensive Care Unit (NICU) were randomly allocated to NIPPV and CPAP. Outcomes of respiratory support were observed and information on risk factors were obtained by going through bed head ticket.

DETAILED DESCRIPTION:
Objective of the study:

To compare the effectiveness of CPAP and NIPPV in neonates with mild to moderate respiratory distress.

Specific objectives To determine the effectiveness of CPAP and NIPPV in neonates with mild to moderate respiratory distress To describe neonatal factors associated with CPAP and NIPPV support. To compare the length of hospital stay in neonates who received CPAP and NIPPV To compare the time taken to achieve full enteral nutrition in neonates who received CPAP and NIPPV.

Study design:

Randomized controlled trial

Study setting:

Study carried out in NICU of the Sri Jayawardanapura General Hospital There are 06 ventilators in NICU of Sri Jayawardanapura Hospital. (Three SLE 2000 infant ventilators and three Bear CUB 750 psv infant ventilators.) Respiratory support (conventional ventilation, CPAP and NIPPV) gave through these ventilators. The neonatal soft tip curved nasal canula with tubing will be use for non invasive respiratory support. The nasal canula connected to the ventilator via an endotracheal tube connector. Systems were regularly monitored. Canula size was chosen to comfortably fit the infant's nostrils.

CPAP started with Positive end expiratory pressure (PEEP) 05 and increased up to PEEP 09 according to the severity of baby's condition.

NIPPV started with intermittent Mandatory ventilation (IMV) rate 30, peak inspiratory pressure (PIP) 20 and PEEP 5.Increased the settings according to the severity of baby's condition.

Sampling Method. All neonates fulfilling inclusion and exclusion criteria registered in the study. And a serial number issued. They were allocated to the two arms of study randomly based on a previously generated random allocation schedule.

They were managed according to hospital management protocol and outcome data were collected from the bed head ticket.

The ethical approval taken from the Ethical Review Committee of Sri Jayawardenepura General Hospital kotte.

Approval taken from Medical Technology and supplies sub committee on clinical trials Written informed consent obtained from parents or guardians of eligible infants before randomization The data sheets did not contain the name and be anonymous. Data stored under lock and key with restricted access only to the principal investigators. The computerized data were password protected and is only available to the investigators.

ELIGIBILITY:
Inclusion Criteria:

All neonates with mild to moderate respiratory distress, requiring non invasive respiratory support on admission as defined by one or more of the following

1. Respiratory distress needing 3L of O2 to maintain saturation of >90%
2. Silverman Anderson score of 4 - 6
3. Apnoea

   1. >2 apnoeic attacks needing tactile stimulation for recovery.
   2. One apnoea needs resuscitation

Exclusion Criteria:

1. Major congenital anomalies
2. Presence of cardiovascular instability {sepsis, anemia or severe intraventricular haemorrhage (IVH)}.
3. Intubation needed on admission to the NICU
4. Consent not provided or refused
5. Major cardiac disease (not including patent ductus arteriosus [PDA]),

   -

Ages: 20 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-28 (Actual)

PRIMARY OUTCOMES:
Non invasive respiratory support failure | 72 hours
  Failure of non invasive respiratory support by requirement for endotracheal ventilation with in 72 hours of starting treatment.

SECONDARY OUTCOMES:
duration of respiratory support | 21 days
  Time in days to stop oxygen support and the neonate to be on room air without respiratory distress or apnoea.
length of hospital stay | 28 days
  The total duration of hospital stay in days.
Grade III and IV Intra Ventricular Haemorrhage (IVH) | 14 days
  Evidence of grade III or IV IVH from ultrasound scan of the brain.
time taken to achieve full enteral nutrition | 21 days
  Total time in days the neonate will receive total enteral feed without intravenous fluid.

CONTACTS AND LOCATIONS:
Overall Officials: ANNE KS GOMEZ, MBBS,MD, Principal Investigator — Teaching Hospital Mahamodara
Locations (1):
- Sri Jayawardanapura teaching hospital, Colombo, Western Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DK Guha, editors, Jaypee Brothers. NNF Recommended Basic Perinatal-Neonatal Nomenclature. Neonatology- Principles and Practice. 1st ed. New Delhi, 1998: 131-2
- [Background] J Crowther ANNP Updated by Dr Smith. East Cheshire NHS trust Endotracheal Intubation guide line February 2013 Version 2.0 3
- [Background] Bhandari V. Nasal intermittent positive pressure ventilation in the newborn: review of literature and evidence-based guidelines. J Perinatol. 2010 Aug;30(8):505-12. doi: 10.1038/jp.2009.165. Epub 2009 Oct 22. PMID 19847188
- [Background] Perinatal society of Sri Lanka in collaborating with WHO collaborating centre for training and research in new born care, All India Institute of Medical Science.Work book on neonatal ventilation.Learner's guide April 2008.
- [Result] Khalaf MN, Brodsky N, Hurley J, Bhandari V. A prospective randomized, controlled trial comparing synchronized nasal intermittent positive pressure ventilation versus nasal continuous positive airway pressure as modes of extubation. Pediatrics. 2001 Jul;108(1):13-7. doi: 10.1542/peds.108.1.13. PMID 11433048
- [Result] Santin R, Brodsky N, Bhandari V. A prospective observational pilot study of synchronized nasal intermittent positive pressure ventilation (SNIPPV) as a primary mode of ventilation in infants > or = 28 weeks with respiratory distress syndrome (RDS). J Perinatol. 2004 Aug;24(8):487-93. doi: 10.1038/sj.jp.7211131. PMID 15141265
- [Result] Lin CH, Wang ST, Lin YJ, Yeh TF. Efficacy of nasal intermittent positive pressure ventilation in treating apnea of prematurity. Pediatr Pulmonol. 1998 Nov;26(5):349-53. doi: 10.1002/(sici)1099-0496(199811)26:53.0.co;2-7. PMID 9859905
- [Result] Barrington KJ, Bull D, Finer NN. Randomized trial of nasal synchronized intermittent mandatory ventilation compared with continuous positive airway pressure after extubation of very low birth weight infants. Pediatrics. 2001 Apr;107(4):638-41. doi: 10.1542/peds.107.4.638. PMID 11335736
- [Result] De Paoli AG, Davis PG, Lemyre B. Nasal continuous positive airway pressure versus nasal intermittent positive pressure ventilation for preterm neonates: a systematic review and meta-analysis. Acta Paediatr. 2003;92(1):70-5. doi: 10.1111/j.1651-2227.2003.tb00472.x. PMID 12650303
- [Result] Lemyre B, Davis PG, De Paoli AG, Kirpalani H. Nasal intermittent positive pressure ventilation (NIPPV) versus nasal continuous positive airway pressure (NCPAP) for preterm neonates after extubation. Cochrane Database Syst Rev. 2017 Feb 1;2(2):CD003212. doi: 10.1002/14651858.CD003212.pub3. PMID 28146296
- [Result] Meneses J, Bhandari V, Alves JG, Herrmann D. Noninvasive ventilation for respiratory distress syndrome: a randomized controlled trial. Pediatrics. 2011 Feb;127(2):300-7. doi: 10.1542/peds.2010-0922. Epub 2011 Jan 24. PMID 21262883
- [Result] Sai Sunil Kishore M, Dutta S, Kumar P. Early nasal intermittent positive pressure ventilation versus continuous positive airway pressure for respiratory distress syndrome. Acta Paediatr. 2009 Sep;98(9):1412-5. doi: 10.1111/j.1651-2227.2009.01348.x. Epub 2009 Jun 12. PMID 19523049
- [Result] Meneses J, Bhandari V, Alves JG. Nasal intermittent positive-pressure ventilation vs nasal continuous positive airway pressure for preterm infants with respiratory distress syndrome: a systematic review and meta-analysis. Arch Pediatr Adolesc Med. 2012 Apr;166(4):372-6. doi: 10.1001/archpediatrics.2011.1142. PMID 22474063
- [Result] Roberts CT, Davis PG, Owen LS. Neonatal non-invasive respiratory support: synchronised NIPPV, non-synchronised NIPPV or bi-level CPAP: what is the evidence in 2013? Neonatology. 2013;104(3):203-9. doi: 10.1159/000353448. Epub 2013 Aug 28. PMID 23989138
- [Result] Claure N, Bancalari E. New modes of mechanical ventilation in the preterm newborn: evidence of benefit. Arch Dis Child Fetal Neonatal Ed. 2007 Nov;92(6):F508-12. doi: 10.1136/adc.2006.108852. Epub 2007 Sep 5. No abstract available. PMID 17804519
- [Result] Kugelman A, Feferkorn I, Riskin A, Chistyakov I, Kaufman B, Bader D. Nasal intermittent mandatory ventilation versus nasal continuous positive airway pressure for respiratory distress syndrome: a randomized, controlled, prospective study. J Pediatr. 2007 May;150(5):521-6, 526.e1. doi: 10.1016/j.jpeds.2007.01.032. PMID 17452229
- [Result] Lemyre B, Laughon M, Bose C, Davis PG. Early nasal intermittent positive pressure ventilation (NIPPV) versus early nasal continuous positive airway pressure (NCPAP) for preterm infants. Cochrane Database Syst Rev. 2016 Dec 15;12(12):CD005384. doi: 10.1002/14651858.CD005384.pub2. PMID 27976361
- [Result] Bisceglia M, Belcastro A, Poerio V, Raimondi F, Mesuraca L, Crugliano C, Corapi UP. A comparison of nasal intermittent versus continuous positive pressure delivery for the treatment of moderate respiratory syndrome in preterm infants. Minerva Pediatr. 2007 Apr;59(2):91-5. PMID 17404558
- [Result] Ramanathan R, Sekar KC, Rasmussen M, Bhatia J, Soll RF. Nasal intermittent positive pressure ventilation after surfactant treatment for respiratory distress syndrome in preterm infants <30 weeks' gestation: a randomized, controlled trial. J Perinatol. 2012 May;32(5):336-43. doi: 10.1038/jp.2012.1. Epub 2012 Feb 2. PMID 22301528
- [Result] Armanian AM, Badiee Z, Heidari G, Feizi A, Salehimehr N. Initial Treatment of Respiratory Distress Syndrome with Nasal Intermittent Mandatory Ventilation versus Nasal Continuous Positive Airway Pressure: A Randomized Controlled Trial. Int J Prev Med. 2014 Dec;5(12):1543-51. PMID 25709790
- [Result] Wood FE, Gupta S, Tin W, Sinha S. Randomised controlled trial of synchronised intermittent positive airway pressure (SiPAP) versus continuous positive airway pressure (CPAP) as a primary mode of respiratory support in preterm infants with respiratory distress syndrome. Archives of Disease in Childhood 2013;98(Suppl 1):A1-117.
- [Result] Lista G, Castoldi F, Fontana P, Daniele I, Cavigioli F, Rossi S, Mancuso D, Reali R. Nasal continuous positive airway pressure (CPAP) versus bi-level nasal CPAP in preterm babies with respiratory distress syndrome: a randomised control trial. Arch Dis Child Fetal Neonatal Ed. 2010 Mar;95(2):F85-9. doi: 10.1136/adc.2009.169219. Epub 2009 Nov 29. PMID 19948523
- [Result] Friedlich P, Lecart C, Posen R, Ramicone E, Chan L, Ramanathan R. A randomized trial of nasopharyngeal-synchronized intermittent mandatory ventilation versus nasopharyngeal continuous positive airway pressure in very low birth weight infants after extubation. J Perinatol. 1999 Sep;19(6 Pt 1):413-8. doi: 10.1038/sj.jp.7200205. PMID 10685270
- [Result] Jasani B, Nanavati R, Kabra N, Rajdeo S, Bhandari V. Comparison of non-synchronized nasal intermittent positive pressure ventilation versus nasal continuous positive airway pressure as post-extubation respiratory support in preterm infants with respiratory distress syndrome: a randomized controlled trial. J Matern Fetal Neonatal Med. 2016;29(10):1546-51. doi: 10.3109/14767058.2015.1059809. Epub 2015 Jul 28. PMID 26135774
- See also: Mechanical ventilation in neonates.Version 19.3 — https://www.uptodate.com